CLINICAL TRIAL: NCT03295929
Title: 3D Finite Element Model of Posterior Membranous Labyrinth From in Vivo MRI of Human Temporal Bone
Brief Title: 3D Model of Posterior Membranous Labyrinth of the Inner Ear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6815
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2017-09

CONDITIONS: Reconstruction of the Posterior Membranous Labyrinth
Keywords: 3D model; Inner ear

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this work is to create a three-dimensional (3D) finite element model (FEM) of the human posterior membranous labyrinth, based on in vivo inner ear magnetic resonance imaging (MRI). This model has a pedagogical interest, and can serve as a basis for reflection in cases of atypical benign paroxysmal positional vertigos. It can also serve for mechanical studies of vestibular physiology.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Adult who has performed an imaging of the inner ear

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult who has performed an imaging of the inner ear
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Measure of dimensions of the model to study the validity of the geometry | Creation of 3D model: 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Orl Et de Chirurgie Cervico-Faciale, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No